CLINICAL TRIAL: NCT06902181
Title: Observation of Inhalation of CXMCI-01 Essential Oil on Patients With Mild Cognitive Impairment
Acronym: CXMCI-01-MCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CMUH113-REC1-180
Record Dates: First submitted 2025-03-16; First posted 2025-03-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; aromatherapy; essential oil,; neuroinflammation; neuroprotection; olfactory training
MeSH Terms: conditions — Cognitive Dysfunction; Neuroinflammatory Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group - 100% CXMCI-01 Essential Oil (Experimental): Experimental Group - 100% CXMCI-01 Essential Oil. Used by inhalation in the morning and night.
  Interventions: Behavioral: Experimental Group - 100% CXMCI-01 Essential Oil
- Control Group - 0.1% CXMCI-01 Essential Oil (placebo) (Placebo Comparator): Control Group - 0.1% CXMCI-01 Essential Oil (Placebo). Used by inhalation in the morning and night.
  Interventions: Behavioral: Control Group - 0.1% CXMCI-01 Essential Oil (placebo)

INTERVENTIONS:
Behavioral: Experimental Group - 100% CXMCI-01 Essential Oil — Participants in the experimental group will inhale 100% CXMCI-01 essential oil twice(CXMCI-01-M in morning, CXMCI-01-N in night) daily for 28 days using an aroma necklace. Each session involves placing 2 drops of the essential oil on a cotton pad inside the necklace. Inhale near the nose for 5 minutes, then wear the aroma necklace and continue inhalation for 60 minutes.
  Arms: Experimental Group - 100% CXMCI-01 Essential Oil
Behavioral: Control Group - 0.1% CXMCI-01 Essential Oil (placebo) — Participants in the placebo group will inhale a 0.1% CXMCI-01 essential oil dilution twice (CXMCI-01-M in morning, CXMCI-01-N in night) ) daily for 28 days. The protocol mirrors the experimental group: inhalation near the nose for 5 minutes, followed by wearing an aroma necklace infused with the diluted essential oil for 60 minutes. This group serves as a placebo comparator to evaluate the effectiveness of the experimental intervention.
  Arms: Control Group - 0.1% CXMCI-01 Essential Oil (placebo)

SUMMARY:
Memory declined and cognitive impairment are common complaints in neurology clinics. Before diagnosing as dementia, individuals will undergo a transition period, including mild cognitive impairment (MCI). Neuroinflammation is an important mechanism of memory problems. For patients with MCI, there are limited available medications. Currently, there is no standardized treatment in Taiwan. The purpose of this study is to explore alternative treatment with essential oil by inhalation to improve memory, sleep, mood, and quality of life for patients with MCI.

This study will include patients who are clinically diagnosed as MCI by a neurologist. This is a double-blind randomized controlled trial, which will include 100 participants with 1:1 allocation into the intervention group and control group. The experimental group will receive 100% CXMCI-01-M Essential Oil every morning and 100% CXMCI-01-N Essential Oil by inhalation every night. The control group will receive 0.1% CXMCI-01-M Essential Oil every morning and 0.1% CXMCI-01-N Essential Oil by inhalation every night. The intervention method involves inhaling for 5 minutes, followed by wearing an essential oil necklace for 60 minutes. Examinations will be conducted before intervention (first visit, V1) and 28 days later (second visit, V2). After 28 days of finishing intervention, the third visit (V3) will be conducted. The primary outcome is the Contextual Memory Test (CMT). Secondary outcomes are Montreal Cognitive Assessment (MoCA), Taiwan Odd-Even Number Sequencing Test (TOENST), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), Pittsburgh Sleep Quality Index (PSQI), and 36-Item Short Form Health Survey (SF-36). Serum biomarkers of amyloid, tau protein, and metabolomics will be checked, as well as urine biomarkers related to neuroinflammation, including lipid peroxidation (LPO), 8-hydroxy-2-deoxyguanosine (8-OHdG), kynurenine, picolinate, quinolinate, and kynurenate. Changes in meridian energy will also be examined by M.E.A.D. and HRV before and after the intervention. It is expected that this study will contribute to the clinical application of CXMCI-01 Essential Oil in patients with MCI and improve their memory, mood, and sleep quality.

DETAILED DESCRIPTION:
< Trial Description and Rationale for Intervention >

Neurodegenerative diseases such as Alzheimer's disease (AD), Parkinson's disease (PD), Lewy body dementia (LBD), and frontotemporal dementia (FTD) are major causes of cognitive decline, with AD being the most prevalent. Dementia is characterized by cognitive impairment, memory deficits, and neuropsychiatric symptoms, leading to loss of independence and increased caregiver burden. Current pharmacological treatments can only slow disease progression, with no curative therapy available.

The pathogenesis of neurodegeneration involves multiple mechanisms, including amyloid-beta (Aβ) aggregation, tau protein hyperphosphorylation, neuroinflammation, oxidative stress, and cholinergic dysfunction. Neuroinflammation, primarily mediated by microglia and astrocytes, plays a central role in neuronal damage. Dysregulated microglia contribute to synaptic dysfunction, while pro-inflammatory astrocytes promote neuronal apoptosis through the NF-κB pathway. Oxidative stress exacerbates neurodegeneration by inducing mitochondrial dysfunction and increasing reactive oxygen species (ROS), which further promote Aβ accumulation and tau pathology.

Mild cognitive impairment (MCI) represents an intermediate stage between normal cognition and dementia. Approximately 25 percent of individuals with MCI progress to dementia within two years, while others may recover cognitive function. Current interventions, including cholinesterase inhibitors, dietary supplements, and exercise, have shown inconsistent results. Given the multifactorial nature of MCI and the potential for cognitive recovery, exploring alternative neuroprotective therapies is essential.

Olfactory dysfunction is an early biomarker of neurodegeneration, as the olfactory nerve directly connects to the limbic system, which regulates memory and emotion. Aromatherapy, the therapeutic use of essential oils, has been investigated for its effects on cognitive function. Studies on cellular and animal models have demonstrated that essential oils exert neuroprotective effects through multiple mechanisms, including reducing Aβ-induced neurotoxicity, modulating microglia-mediated neuroinflammation, regulating glutamate and GABA neurotransmission, and inhibiting tau hyperphosphorylation via glycogen synthase kinase-3β (GSK3β) suppression. Essential oils also activate cAMP response element-binding protein (CREB) signaling, enhance antioxidant defense by increasing superoxide dismutase (SOD) levels, reduce pro-inflammatory cytokines such as TNF-α, IL-1β, and IL-6, and modulate brain-derived neurotrophic factor (BDNF) expression. Additionally, they prevent neuronal apoptosis and mitochondrial dysfunction, inhibit acetylcholinesterase (AChE) activity, and enhance synaptic plasticity and neurotransmitter balance.

Several essential oil constituents, including 1,8-cineole, linalool, limonene, thymol, alpha-humulene, cis-carveol, alpha-pinene, beta-pinene, rosmarinic acid, and zingerone, have demonstrated neuroprotective properties. These compounds may contribute to cognitive enhancement by reducing neuroinflammation, oxidative stress, and synaptic dysfunction.

Based on this hypothesis, the investigators formulated a natural essential oil blend rich in 1,8-cineole, linalool, limonene, and other bioactive compounds, and applied it via inhalation as an intervention. Using the concept of olfactory training and targeting the limbic system, the study aims to evaluate whether essential oil inhalation can promote improvements in cognition, memory, sleep, mood, and quality of life in individuals with MCI. The effects will be assessed through validated clinical scales and by measuring urine and serum biomarkers related to neuroinflammation. Additionally, changes in meridian energy and autonomic nervous system activity will be monitored. The goal is to provide a convenient and supportive complementary therapy for individuals with MCI, offering clinicians an evidence-based option for early intervention in cognitive decline.

< Study Procedures and Design Rationale>

This study is a randomized, double-blind, parallel-group clinical trial designed to evaluate the effects of CXMCI-01 essential oil inhalation on cognitive function in individuals with mild cognitive impairment (MCI). A total of 100 participants will be enrolled and randomly allocated in a 1:1 ratio to either the experimental group or the control group.

Randomization will be conducted using a computer-generated sequence, and allocation will be concealed using opaque, sealed envelopes. Each participant will receive a sequential identification number. The randomization process and distribution of the essential oil formulations will be managed by a third party who is independent of the study procedures to ensure blinding.

Participants will be recruited through neurology outpatient clinics at China Medical University Hospital, Chung Shan Medical University Hospital, and Everan Hospital. Those who meet preliminary eligibility will undergo final screening and informed consent at Everan Hospital.

The study consists of three scheduled visits:

* Visit 1 (V1): Baseline assessment prior to intervention.
* Visit 2 (V2): Post-intervention assessment after 28 days of essential oil inhalation. A visit window of + 5 days from the scheduled date is acceptable.
* Visit 3 (V3): Follow-up assessment conducted 28 days after the completion of the observation period. A visit window of ±5 days is also acceptable.

The essential oil intervention includes two types of blended formulations, each prepared in two concentrations (100% and 0.1%):

* CXMCI-01-M: A blend containing lemon, rosemary (1,8-cineole type), rose geranium, and sweet marjoram essential oils.
* CXMCI-01-N: A blend containing frankincense, true lavender, linalool, and ylang-ylang essential oils.
* The control group are diluted to 0.1% concentration using a neutral carrier oil.

Participants will perform inhalation twice daily for 28 consecutive days. And use twice daily. The essential oil intervention was designed with consideration of the body's natural circadian rhythm. The autonomic nervous system exhibits daily fluctuations, with sympathetic activity typically dominant in the morning and parasympathetic activity more prominent at night. Cortisol levels also follow a diurnal pattern, peaking in the early morning and gradually declining throughout the day. To align with this physiological rhythm, the morning formulation (CXMCI-01-M) was selected to support alertness and sympathetic activation, while the evening formulation (CXMCI-01-N) was intended to promote relaxation and enhance parasympathetic activity. This time-specific approach aims to optimize the neurophysiological effects of essential oil inhalation, supporting both cognitive performance and overall well-being.

* In the morning, 2 drops of the assigned essential oil (intervention group with 100% formula, placebo group with 0.1% formula) will be applied to a cotton pad. Participants will first inhale the aroma near the nose for 5 minutes before placing the cotton pad in an aroma necklace, which will be worn for an additional 60 minutes.
* The same procedure will be repeated at night with a different formulation.

The experimental group will receive the 100% CXMCI-01 formulations (CXMCI-01-M in the morning and CXMCI-01-N at night), while the control group will receive the 0.1% diluted versions of the same formulas.

To ensure consistency, participants will be instructed to avoid interfering factors during inhalation, such as eating, drinking strong-smelling beverages, smoking, or being in scented environments. Concurrent use of other essential oils, perfumes, or cognitive-enhancing treatments will be restricted throughout the study period.

This structured inhalation protocol, utilizing specific essential oil compositions with known neuroprotective properties, is designed to target neuroinflammatory and oxidative mechanisms through the olfactory-limbic pathway. The study aims to explore whether this intervention can support cognitive, emotional, and physiological well-being in patients with MCI.

Throughout the study period, participants or their caregivers will be asked to maintain a daily log, recording aromatherapy usage, sleep patterns (including bedtime, time to fall asleep, and wake-up time), physical activity (type and duration), and dietary habits. Specific attention will be given to the intake of refined sweets, sugary beverages, and fried or grilled foods. Participants will also document any acute medical events, such as hospital visits, medication use, and symptoms of upper respiratory infections. Any adverse reactions potentially related to essential oil use, such as dizziness, palpitations, or asthma-like symptoms, will be reported in the log.

Following the post-intervention assessment, participants will continue to maintain their daily tracking logs as previously instructed. A follow-up evaluation will be conducted within 28 ± 5 days after the completion of the intervention to examine the sustained effects of the essential oil inhalation.

The follow-up assessments will include a combination of clinical, cognitive, psychological, and physiological evaluations. Cognitive assessments will include the Contextual Memory Test (CMT), a standardized tool for assessing episodic memory in real-life contexts; the Montreal Cognitive Assessment (MoCA), commonly used to screen for mild cognitive impairment; and the Taiwan Odd-Even Number Sequencing Test (TOENST), which evaluates working memory and processing speed.

Psychological and quality of life assessments will include the Pittsburgh Sleep Quality Index (PSQI), Beck Depression Inventory (BDI), Beck Anxiety Inventory (BAI), and the 36-Item Short Form Health Survey (SF-36), which collectively assess sleep quality, emotional well-being, and overall health-related quality of life.

To explore the potential biological effects of the essential oil intervention, blood samples will be collected for biomarker analysis. These may include markers related to amyloid and tau protein pathways, such as the Aβ42/40 ratio, total tau protein, and phosphorylated tau protein-217 (p-tau 217), which are commonly associated with neurodegenerative processes and Alzheimer's disease pathology. Including these biomarkers will allow for an exploratory evaluation of possible changes in biological mechanisms relevant to cognitive decline and mild cognitive impairment.

In addition to blood-based markers, urinary biomarkers related to neuroinflammation will also be assessed at baseline and post-intervention. These may include lipid peroxidation (LPO) and 8-hydroxy-2-deoxyguanosine (8-OHdG), quinolinate, kynurenine, kynurenate, and picolinate. These biomarkers are involved in oxidative stress, mitochondrial function, and neuroimmune activity, and may provide further insights into the systemic biological response to the intervention.

Physiological assessments will include non-invasive testing using the Meridian Energy Analysis Device (M.E.A.D.) to evaluate meridian energy distribution, and heart rate variability (HRV) testing to assess autonomic nervous system function. These comprehensive follow-up evaluations aim to assess the longer-term impact of CXMCI-01 essential oil inhalation on cognitive function, emotional status, sleep quality, biological markers of neuroinflammation and neurodegeneration, and systemic physiological regulation.

To minimize variability, participants will follow dietary and lifestyle restrictions before each testing session. This includes avoiding excessive oily food and refined carbohydrates for three days before testing and refraining from alcohol or caffeinated beverages the day before. Morning urine samples will be collected on scheduled days, and female participants will be asked to avoid urine collection during menstruation.

This comprehensive assessment protocol aims to evaluate not only cognitive changes but also neuroinflammatory markers, autonomic nervous system function, and energy regulation in response to essential oil inhalation.

< Study Summary and Expected Impact >

This randomized, double-blind, parallel-group trial is designed to evaluate the effects of CXMCI-01 essential oil inhalation on cognitive function in individuals with mild cognitive impairment (MCI). By integrating daily olfactory stimulation based on circadian rhythm, this study aims to explore whether specific essential oil formulations can influence neuroinflammation, oxidative stress, and autonomic function to support cognitive health.

Through a comprehensive multimodal assessment, including cognitive evaluations, biomarker analysis, and physiological testing, this study will generate valuable data on the potential of essential oil-based interventions as a complementary approach to MCI management. The findings may contribute to future clinical applications by providing an evidence-based strategy for cognitive enhancement and neuroprotection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50 years or older, presenting with memory and cognitive impairment. Diagnosed with Mild Cognitive Impairment (MCI) by a neurologist based on clinical and psychological assessment. Mini-mental state examination(MMSE) ≥ 23 and Clinical Dementia Rating (CDR) = 0.5.
2. Neurological consultation: Participants must undergo a neurology consultation, including medical history review, neurological examination, and olfactory function testing.
3. No essential oil use within the past month.

Exclusion Criteria:

1. Dementia caused by other conditions, including: Alzheimer's disease, Parkinson's disease, vascular dementia, traumatic brain injury, central nervous system infections or multiple sclerosis
2. Cognitive impairment due to brain lesions, such as: brain tumors, hydrocephalus, severe brain atrophy
3. Severe metabolic disorders potentially affecting cognitive function, including:

   1. Uncontrolled hyperthyroidism or hypothyroidism
   2. Uncorrected electrolyte imbalance
   3. Liver dysfunction (ALT or AST > 1.5× normal upper limit)
   4. Renal dysfunction (Creatinine > 1.5× normal upper limit)
   5. Uncontrolled or poorly managed diabetes (Random glucose > 200 mg/dL and HbA1c > 8%)
   6. Uncontrolled or poorly managed hypertension (SBP > 160 mmHg or DBP > 100 mmHg)
   7. Uncorrected vitamin B12 or folate deficiency
   8. Severe anemia (Hb < 8 g/dL) or acute bleeding causing Hb < 8 g/dL
   9. Current severe infection (fever > 38°C, ongoing antibiotic use, or abnormal WBC count)
   10. Body Mass Index (BMI) ≥ 35
4. Severe nasal or pharyngeal diseases affecting olfactory function, or history of asthma attacks in the past six months.
5. Substance or alcohol abuse within the past two years, meeting DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) criteria.
6. Diagnosis of psychiatric disorders within the past year, including: Major depressive disorder, schizophrenia, bipolar disorder (DSM-5 criteria),
7. Severe insomnia, defined as:

(1) Experiencing insomnia symptoms for more than 50% of days per month for at least three months, causing daytime fatigue.

(2) Use of three or more sleep-related medications (e.g., benzodiazepines or Z-drugs).

8. History of cancer under active treatment. 9. Use of anticholinergic or acetylcholinesterase inhibitor medications. 10.Concurrent use of other neuroprotective therapies, including traditional Chinese medicine or dietary supplements (except for long-term users exceeding three months).

11.Allergy to essential oils. 12.Inability to comply with essential oil inhalation procedures. 13.Other conditions deemed inappropriate by the principal investigator. 14.Inability to understand or comply with study procedures, or failure to sign the informed consent form.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Contextual Memory Test (CMT) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Contextual Memory Test (CMT) is a standardized cognitive assessment used to evaluate memory function in individuals with mild cognitive impairment (MCI). The test measures both immediate and delayed recall of visual stimuli in a structured context. At each study visit, participants will complete both immediate and delayed recall tasks. Each section is scored out of 20 points, resulting in a total raw score ranging from 0 to 40. Higher scores indicate better memory performance. This assessment provides a quantitative and repeatable measure of episodic memory, allowing for longitudinal tracking of cognitive changes throughout the study.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment(MoCA) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Montreal Cognitive Assessment (MoCA) is a widely used cognitive screening tool designed to detect mild cognitive impairment (MCI) and early cognitive decline. It evaluates multiple cognitive domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The total score ranges from 0 to 30, with higher scores indicating better cognitive function. A score of 26 or above is generally considered within the normal range. In this study, the MoCA will be administered at each study visit to assess changes in global cognitive performance over time. The test provides a sensitive and standardized measure for monitoring cognitive outcomes in individuals with MCI.
Taiwan Odd-Even Number Sequencing Test (TOENST) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Taiwan Odd-Even Number Sequencing Test (TOENST) assesses working memory, attention, and executive function by requiring participants to reorganize spoken numbers-placing even numbers in ascending order and odd numbers in descending order. The test consists of seven levels, with each level containing three attempts. The total score ranges from 0 to 21, with higher scores indicating better cognitive performance. If a participant fails all three attempts in a level, the test is discontinued. TOENST will be administered at baseline and follow-up visits to assess changes in cognitive function in individuals with mild cognitive impairment (MCI).
Beck Depression Inventory (BDI) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Beck Depression Inventory (BDI) is a self-report questionnaire designed to assess the severity of depressive symptoms. It consists of 21 items, each rated on a 0 to 3 scale, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms. Score interpretations are generally categorized as minimal (0-13), mild (14-19), moderate (20-28), and severe (29-63). In this study, the BDI will be administered at multiple time points to monitor changes in participants' emotional well-being and track potential improvements or worsening of depressive symptoms during the intervention period.
Beck Anxiety Inventory (BAI) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Beck Anxiety Inventory (BAI) is a 21-item self-report scale developed to assess the severity of anxiety symptoms. Each item is rated on a 0 to 3 scale, with total scores ranging from 0 to 63. Higher scores indicate more severe anxiety. The BAI evaluates symptoms such as nervousness, dizziness, inability to relax, and fear of losing control. Score ranges are commonly interpreted as minimal (0-7), mild (8-15), moderate (16-25), and severe (26-63). In this study, the BAI will be used to assess anxiety levels at baseline and post-intervention to evaluate the emotional effects of the essential oil inhalation program.
Pittsburgh Sleep Quality Index (PSQI) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire designed to assess sleep quality and disturbances over a one-month period. It consists of 19 items covering seven domains, including subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A score above 5 is typically used to identify individuals with significant sleep disturbances.
36-Item Short Form Health Survey (SF-36) | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  The 36-Item Short Form Health Survey (SF-36) assesses health-related quality of life (HRQoL) across eight domains, including physical functioning, pain, general health, vitality, social functioning, and mental health. Scores range from 0 to 100, with higher scores indicating better health status. It provides Physical (PCS) and Mental (MCS) Component Summary scores. The SF-36 will be administered at baseline and follow-up visits to evaluate changes in physical and mental well-being in individuals with mild cognitive impairment (MCI).
Plasma biomarkers related to amyloid and tau pathology | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  Plasma biomarkers related to neurodegeneration and cognitive decline will be assessed. These may include amyloid and tau-related proteins, such as the Aβ42/40 ratio, total tau, and phosphorylated tau (p-tau 217). Biomarker levels will be analyzed based on standard laboratory reference ranges to evaluate their association with mild cognitive impairment (MCI) and potential changes following intervention.
Urinary biomarkers related to oxidative stress and neuroinflammation | Baseline (V1), Post-Intervention (Day 28) (V2)
  Urinary biomarkers will be assessed at baseline and post-intervention to evaluate systemic changes related to oxidative stress and neuroinflammation in individuals with mild cognitive impairment (MCI). Biomarkers of oxidative stress may include lipid peroxidation (LPO) and 8-hydroxy-2-deoxyguanosine (8-OHdG), which reflect redox imbalance and oxidative DNA damage. Neuroinflammation-related biomarkers may include quinolinate, kynurenine, kynurenate, and picolinate, which are metabolites within the kynurenine pathway and are associated with neuroimmune regulation and inflammatory responses. These urine-based markers provide a non-invasive approach to monitoring physiological changes linked to cognitive decline and the potential impact of the intervention.
Meridian energy assessment using M.E.A.D device | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  Meridian energy will be assessed using the Meridian Energy Analysis Device (MEAD) at baseline and post-intervention to evaluate changes in systemic bioenergetic status. The MEAD is a non-invasive tool based on Traditional Chinese Medicine (TCM) principles and operates by measuring electrical conductivity at specific acupoints along the 12 primary meridians. By applying a mild electrical current, the device detects skin resistance and calculates conductivity levels, which reflect the flow and balance of energy (Qi) within each meridian. Variations in conductivity may be associated with autonomic nervous system function, organ system imbalance, or stress-related physiological changes. This assessment will help determine whether the intervention modulates meridian energy patterns in individuals with mild cognitive impairment (MCI).
Heart rate variability (HRV) assessment | Baseline (V1), Post-Intervention (Day 28) (V2), and Follow-up (Day 56) (V3).
  Heart rate variability (HRV) will be measured at baseline and post-intervention to assess autonomic nervous system activity. HRV refers to the variation in time intervals between consecutive heartbeats and is widely used as a non-invasive indicator of sympathetic and parasympathetic nervous system balance. Higher HRV generally reflects greater parasympathetic (vagal) activity and better adaptability to physiological stress, while lower HRV may be associated with stress, fatigue, or dysregulation of autonomic function. In this study, HRV analysis will be used to explore whether the intervention modulates autonomic regulation in individuals with mild cognitive impairment (MCI). Measurements will be taken under resting conditions to ensure consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Huei Liu, NTU, Ph.D. (Biochem & Mol Bio), Principal Investigator — Graduate Institute of Integrated Medicine, China Medical University
Locations (1):
- Everan Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared to protect participant privacy and confidentiality. Due to ethical considerations and data protection regulations, all collected data will be securely stored and used solely for research purposes within the study team.